CLINICAL TRIAL: NCT03712969
Title: Shenlingcao Oral Liquid for Patients With Stage II or IIIA Non-small Cell Lung Cancer Receiving Radical Resection: A Pragmatic, Multicenter Randomized Controlled Trial
Brief Title: Shenlingcao Oral Liquid for Patients With Stage II or IIIA NSCLC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Sun Xin, Director, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20181009
Record Dates: First submitted 2018-10-09; First posted 2018-10-19 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Chemotherapy, Adjuvant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients receive Shenlingcao oral liquid combined with conventional adjuvant chemotherapy, which take 4 courses, 30 days per course, one bottle per day.
  Interventions: Drug: Shenlingcao Oral Liquid
- Control group (No Intervention): Patients receive conventional adjuvant chemotherapy.

INTERVENTIONS:
Drug: Shenlingcao Oral Liquid — Patients receive Shenlingcao oral liquid combined with conventional adjuvant chemotherapy, which take 4 courses, 30 days per course, one bottle per day.
  Arms: Intervention group

SUMMARY:
In this study, a pragmatic, open labelled, multi-center randomized controlled trial will be conducted. The study population are stage II and IIIA NSCLC patients undergoing R0 resection and will be scheduled for adjuvant chemotherapy. Potentially eligible patients will be screened by the research clinicians and requested to complete and sign a consent form before enrolment. Eligible patients who consent to participate will be randomly assigned to the intervention group (patients receive conventional treatment and Shenlingcao oral liquid) and the control group (patients only receive conventional treatment) designed dynamic stratified block randomized algorithm via a central randomization system for clinical research using 1:1 ratio.

The intervention and control group will be enrolled before the first chemoradiation. Non-allelic follow-up will be conducted in this study and terminated when the last enrolled patient follow up to 24 months. Prospectively collected information from patients, including baseline, chemoradiation, use of Shenlingcao Oral Liquid and the other complementary drugs, and various outcome measures (the questionnaire of EORTC QLQ, death, tumor recurrence, tumor metastasis, and chemotherapy-induced side effects of the blood system, etc.). Follow-up points included: Baseline (before giving chemotherapy), 2-3 days after each chemotherapy cycle, and 6,12,18,24,30,36 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older;
* Pathological diagnosis of patients with stage II, III A primary NSCLC;
* R0 resection has been accepted;
* Received adjuvant chemotherapy or adjuvant chemotherapy for the first time after surgery;
* Informed consent has been signed.

Exclusion Criteria:

* Incorporation of other malignant tumors (such as leukemia, liver cancer, etc.);
* Patients with unclear pathological types;
* Patients with unclear pathological staging;
* Preserved Shenlingcao Oral Liquid before R0 resection surgery;
* Received immunotherapy or targeted therapy before R0 resection surgery;
* Radiotherapy and chemotherapy before R0 resection surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
The quality of life assessed by Research and Treatment of Cancer Quality of Life Questionnaire | 2-3 days after the fourth chemotherapy cycle
  We investigated the long-term quality of life of postoperative lung cancer patients, utilizing the disease-specific European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ) C30 to assess the quality of life among these patients. The EORTC QLQ-C30 is composed of 9 multi-item scales including 5 functional scales, 3 symptom scales, a global quality-of-life scale, and 6 single-item symptom measures. All the items are scored on a scale of 0 to 100, with a high score on a functional or the global quality-of-life scale representing a high level of functioning or quality of life and a high score on a symptom scale representing a high level of symptoms.

SECONDARY OUTCOMES:
The completion rate of chemotherapy | 2-3 days after the fourth chemotherapy cycle
  Whether the patient completed four cycles of chemotherapy.
Disease-free survival | 24 months after enrollment
  Disease-free survival (DFS) refers to the time from the operation to the time that there is evidence of tumor recurrence / metastasis or any cause of death (the DFS of lost follow-up patients is the last follow-up time). The tumor recurrence / metastasis needs to be diagnosed based on imaging or pathological evidence.
Remission of hematological toxicity caused by chemotherapeutic drugs | 2-3 days after the fourth chemotherapy cycle
  Remission of hematological toxicity caused by chemotherapeutic drugs, using WHO grading of acute and subacute toxicity. Hematological toxicity is observed from four hematological indicators, including hemoglobin, white blood cells, granulocytes and platelets. A 5-grade system of severity levels is recommended for general use: grades 0-4 . The higher the level, the greater the toxic reaction. The most severe of the four indicators is the patient's hematological toxicity level.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, PhD, Study Director — The West China Hospital of Sichuan university
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Luo X, Liu J, Ma Y, Tan J, Wang W, Hu J, Fu X, Xu L, Yu F, Xu S, Ma H, Yu X, You Q, Wang Z, Li L, Zhang X, Sun X. Shenlingcao oral liquid for patients with non-small cell lung cancer receiving adjuvant chemotherapy after radical resection: A multicenter randomized controlled trial. Phytomedicine. 2023 May;113:154723. doi: 10.1016/j.phymed.2023.154723. Epub 2023 Feb 21. PMID 36871476